CLINICAL TRIAL: NCT02322567
Title: Influence of Left Ventricular Diastolic Dysfunction on Graft Function and Postoperative Complication in Patients Undergoing Elective Kidney Transplantation
Brief Title: Left Ventricular Diastolic Dysfunction in Kidney Recipients
Status: Completed | Type: Observational
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Assistant professor, Severance Hospital
Other Study IDs: 4-2014-0808
Record Dates: First submitted 2014-12-09; First posted 2014-12-23 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Medical Records

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LV diastolic dysfunction
  Interventions: Other: medical records
- No LV diastolic dysfunction
  Interventions: Other: medical records

INTERVENTIONS:
Other: medical records — review of medical records

SUMMARY:
The purpose of this study is to examine the relationship between pre-operative LV diastolic function and post-operative complications and kidney function in living-donor kidney transplantation patients.

ELIGIBILITY:
Inclusion Criteria:

* Elective kidney transplantation patients

Exclusion Criteria:

* No data of preoperative echocardiography

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective kidney transplantation patients
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2012-01; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Patients with postoperative cardiovascular complications | 30 days
  acute myocardial infarction, ventricular fibrillation/tachycardia, cardiogenic shock, newly-onset atrial fibrillation, clinical pulmonary edema requiring endotracheal intubation or dialysis

SECONDARY OUTCOMES:
Patients with postoperative pulmonary edema | 30 days
  pulmonary edema by radiological evidence

OTHER OUTCOMES:
Postoperative graft function (graft failure, acute rejection, graft loss, serum creatinine) | 30 days
  graft failure, acute rejection, graft loss, serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Yong Seon Choi, MD, PhD, Principal Investigator — Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Kim EJ, Chang S, Kim SY, Huh KH, Kang S, Choi YS. Predictive Value of Echocardiographic Abnormalities and the Impact of Diastolic Dysfunction on In-hospital Major Cardiovascular Complications after Living Donor Kidney Transplantation. Int J Med Sci. 2016 Jul 18;13(8):620-8. doi: 10.7150/ijms.15745. eCollection 2016. PMID 27499694